CLINICAL TRIAL: NCT01329627
Title: Phase II Feasibility Study of Weekly Paclitaxel Followed by Weekly Doxorubicin Plus Daily Oral Cyclophosphamide for Locally Advanced HER2-Negative Breast Cancer
Brief Title: Feasibility Study of Metronomic Chemotherapy for Locally Advanced HER2-Negative Breast Cancer
Acronym: TAME-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Fundação Faculdade de Medicina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 50/2010 - TAME
Record Dates: First submitted 2010-11-08; First posted 2011-04-06 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Locally Advanced HER2-negative Breast Cancer
MeSH Terms: interventions — Paclitaxel; AC protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel/doxorubicin/cyclophosphamide (Experimental)
  Interventions: Drug: Paclitaxel/doxorubicin/cyclophosphamide

INTERVENTIONS:
Drug: Paclitaxel/doxorubicin/cyclophosphamide — Metronomic chemotherapy as described below:
  1. Paclitaxel 100 mg/m2 once a week for 8 weeks followed by;
  2. Doxorubicin 24 mg/m2 once a week concomitant to oral cyclophosphamide 100 mg/day (fix dose) for 9 weeks.
  Other Names: Metronomic chemotherapy
Drug: Paclitaxel/doxorubicin/cyclophosphamide — Metronomic chemotherapy as described below:
  Paclitaxel 100 mg/m2 once a week for 8 weeks followed by; Doxorubicin 24 mg/m2 once a week concomitant to oral cyclophosphamide 100 mg/day (fix dose) for 9 weeks.
  Other Names: Metronomic chemotherapy

SUMMARY:
The purpose of this study is to determine whether weekly paclitaxel followed by weekly doxorubicin plus daily oral cyclophosphamide without granulocyte colony-stimulating factor (G-CSF) is feasible in the treatment of locally advanced HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced breast cancer diagnosed by guided core biopsy
* T > 2 cm (any N), or any T and node positive (needle biopsy is required)
* Non-metastatic disease assessed by computed tomography and bone scintigraphy
* Histological grade 2 and Ki67 > 15% or
* Histological grade 3 or
* Any triple negative (TN) or
* Inflammatory breast cancer (IBC)
* Normal left ventricular ejection fraction (LVEF)
* HER2-negative disease

Exclusion Criteria:

* Another malignancy within the last 5 years (except curatively treated skin carcinoma, in situ cervix carcinoma, in situ ductal carcinoma of the breast, or in situ lobular carcinoma of the breast)
* Clinically significant comorbidities as cardiovascular diseases, chronic obstructive pulmonary disease (COPD), renal or liver failure, psychiatric disorders
* LVEF value below institutional limits of normal
* Predominant lobular carcinoma histology
* Grade 1 tumors
* Detected or suspicious distant metastasis
* Neutrophils less than 1,500/µL, platelets less than 100,000/µL, hemoglobin less than 10 g/dL, AST more than 2.5x upper limit of normal (ULN), total bilirubin more than ULN, alkaline phosphatase more than 1.5x ULN
* Male sex
* HER2-positive breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia | 18 weeks
  Incidence of febrile neutropenia with modified metronomic schedule (whithout GCSF) will be no higher than 10%

SECONDARY OUTCOMES:
Efficacy | From the beginning of treatment until surgery, progression and death
  Efficacy will be assessed by:
  1. Tumor measurements using MRI
  2. Pathologic complete response
  3. Progression-free survival
  4. Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- State of Sao Paulo Cancer Institute, São Paulo, São Paulo, Brazil